CLINICAL TRIAL: NCT02767817
Title: The Safety and Efficacy Assessment of Injectable Collagen Scaffold™ Combined With Mesenchymal Stem Cells Transplantation in Patients With Brain Injury
Brief Title: Injectable Collagen Scaffold™ Combined With MSCs Transplantation for Brain Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Affiliated Hospital of Logistics University of CAPF (Other)
Responsible Party: Principal Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAS-XDA-BI/IGDB
Record Dates: First submitted 2016-04-29; First posted 2016-05-10 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2016-04

CONDITIONS: Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stereotactic Hematoma Evacuation (Sham Comparator)
  Interventions: Procedure: Stereotactic Hematoma Evacuation
- MSCs Transplantation (Experimental)
  Interventions: Biological: MSCs Transplantation
- Injectable Collagen Scaffold with MSCs Transplantation (Experimental)
  Interventions: Biological: Injectable Collagen Scaffold with MSCs Transplantation

INTERVENTIONS:
Procedure: Stereotactic Hematoma Evacuation — Stereotactic intracranial hematoma and insert the drainage tube to inhale haematoma. The drainage tube stayed in the position for 1-2 days until adequate drainage of hematomas, and then the drainage tube was pulled out.
  Arms: Stereotactic Hematoma Evacuation
Biological: MSCs Transplantation — Stereotactic intracranial hematoma and insert the drainage tube to inhale haematoma. The drainage tube stayed in the position for 1-2 days until adequate drainage of hematomas,and 10 million MSCs were transplanted into the hematoma cavity before the drainage tube was pulled out.
  Arms: MSCs Transplantation
Biological: Injectable Collagen Scaffold with MSCs Transplantation — Stereotactic intracranial hematoma and insert the drainage tube to inhale haematoma. The drainage tube stayed in the position for 1-2 days until adequate drainage of hematomas, and injectable collagen scaffold combined with 10 million MSCs were transplanted into the hematoma cavity before the drainage tube was pulled out.
  Arms: Injectable Collagen Scaffold with MSCs Transplantation

SUMMARY:
The purpose of this study is to assess the safety and efficacy of injectable collagen scaffold combined with Mesenchymal stem cells (MSCs) transplantation in patients with brain injury.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female，35-75 years old.
2. The surgery time should be > 6 hours after symptom onset.
3. Glasgow coma score (GCS) was 9-15.
4. CT diagnosis of intracerebral hemorrhage (25-40 ml), except for patients with signs of craniotomy to remove the hematoma.
5. Signed informed consent obtained from the patient or patient's legally authorized representative.

Exclusion Criteria:

1. Glasgow coma scale of <8.
2. Patients suffering severe heart failure, severe lung disease, uremia, cirrhosis, end-stage cancer, coagulation disorders, stroke sequela.
3. Asphyxia, cardiac arrest or successful cardiopulmonary resuscitation before hospitalization.
4. Lactating or pregnant woman.
5. Refuse to sign informed content.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events and participants with those adverse events | 24 month
  Proportion of patients with postoperative infections and serious adverse events (SAEs) will be assessed by long term follow-up.

SECONDARY OUTCOMES:
Change in functional outcomes as measured by National Institutes of Health stroke scale (NIHSS) score | baseline, day 1-7, and 1, 3, 6, 12, 18 and 24 month after surgery
Change in motor recovery evaluated by Brunnstrom stage | 1, 3, 6, 12, 18 and 24 month after surgery
Change in self-care ability as measured by Barthel Index (BI) | 1, 3, 6, 12, 18 and 24 month after surgery
Change in pain intensity as measured by Visual Analogue Scale (VAS) | 1, 3, 6, 12, 18 and 24 month after surgery
Change in electrical brain activity as measured by Electroencephalography (EEG) | baseline, day 1, 4, 7, and 1, 3, 6, 12, 18, 24 month after surgery
Changes in brain electrophysiology as measured by Somatosensory evoked potential (SSEP) | baseline, day 1,4,7, and 1, 3, 6, 12, 18, 24 month after surgery
Change in brain pathology diagnosed by Head CT scan | baseline, day 1,4,7, and 1, 3, 6, 12, 18, 24 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Ph.D, Principal Investigator — Chinese Academy of Sciences
Locations (1):
- Affiliated Hospital of Logistics Universtiy of CAPF, Tianjin, China